CLINICAL TRIAL: NCT00000569
Title: The Chronic Obstructive Pulmonary Disease Early Intervention Trial
Brief Title: Lung Health Study II
Acronym: LHSII
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 9109M04382; 5U01HL050267-03 (NIH)
Record Dates: First submitted 1999-10-27; First posted 1999-10-28 (Estimated); Last update posted 2019-11-01 (Actual); Status verified 2019-10

CONDITIONS: Lung Diseases; Lung Diseases, Obstructive; Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Lung Diseases; Lung Diseases, Obstructive; Pulmonary Disease, Chronic Obstructive | interventions — Triamcinolone; Triamcinolone Acetonide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Triamcinolone (Active Comparator): 1200 micrograms of triamcinolone in daily divided doses
  Interventions: Drug: triamcinolone
- Placebo (Placebo Comparator): Placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: triamcinolone — 1200 micrograms of triamcinolone in daily divided doses
  Other Names: Azmacort
  Arms: Triamcinolone
Other: Placebo — Placebo
  Arms: Placebo

SUMMARY:
To determine if participants with chronic obstructive pulmonary disease, who were assigned to inhaled corticosteroids had a lower rate of decline in lung function and lower incidence of respiratory morbidity compared to participants assigned to placebo.

DETAILED DESCRIPTION:
BACKGROUND:

Chronic obstructive pulmonary disease (COPD), the fourth leading cause of death in the United States and a major cause of morbidity, is a spectrum of chronic lung diseases including clinical diagnoses of chronic bronchitis, emphysema, and combinations of both. Varying degrees of bronchoreactivity occur over the entire spectrum. Asthma and COPD have many features in common. Distinction is usually dependent on clinical features and clinical course. The diagnosis of asthma will not exclude a patient from the designation of COPD for this study, although criteria for exclusion include recent (within six months) use of inhaled or oral steroid with the intent of excluding most of those who are clearly predominantly bronchospastic. The morbid anatomy of COPD is well described and includes many features of acute and chronic inflammation. There is well supported evidence in the literature that this inflammatory process may be an important pathogenetic mechanism in the development of emphysema. On this basis, the rationale for the use of corticosteroids is well justified. There are various published studies suggesting that inhaled steroids reduce bronchial lavage markers of inflammation, variously influence short-term bronchial hyperreactivity, improve lung function acutely or short-term, and slow rate of decline in lung function. Most studies have asked for improvement rather than stability. However, despite the studies which do not support these contentions and the lack of long-term information, inhaled steroids in COPD are becoming widely used in clinical practice. It was the intent of this clinical trial to assess the long-term efficacy of this treatment before such therapy became an accepted community practice, making it impractical or impossible to conduct a clinical trial.

DESIGN NARRATIVE:

Subjects were recruited from the Lung Health Study I and randomized to 1200 micrograms of triamcinolone in daily divided doses or to placebo. Pulmonary function was evaluated every six months. Bronchial activity was tested at baseline, at nine months, and at three-and-a-half years using a methacholine inhalation challenge. Mean duration of follow-up was 40 months. The primary outcome measure was the rate of decline in pulmonary function as assessed by the post-bronchodilator forced expiratory volume at one second (FEV1) value. Other outcome measures included death, respiratory symptoms, quality of life, side-effects and toxicity, adherence, bronchial hyperreactivity, atopic status, and smoking status. Recruitment was initiated in November 1994 and ended November 28, 1995 to allow 3.5 to 4.5 years of follow-up through April, 1999.

The investigators initiated a dose monitor (puff counter) protocol at nine of the centers among the fair to satisfactory compliers (4 to 9 puffs versus the ideal of 12 puffs per day) to test whether a memory aid would enhance inhaler compliance. Consenting participants were randomized to Group 1 who could see the display on the puff counter for 12 months or to Group 2 who had no counter for three months, a counter that recorded but did not display for three months, and a counter with display for six months.

There were a bone densitometry and adrenal suppression ancillary studies, funded by Rhone-Poulenc-Rorer, to assess the effect of inhaled corticosteroids on bone density and adrenal function.

ELIGIBILITY:
Inclusion:

1. Previously participated in or screened for the Lung Health Study I
2. Ages 40 to 69
3. Forced expiratory volume at one second (FEV1)/forced vital capacity(FVC) < 70 percent
4. Forced expiratory volume at one second (FEV1) 30 to 90 percent predicted.

Exclusions:

1. Cancer
2. Recent myocardial infarction
3. Alcoholism
4. Heart Failure
5. Insulin-dependent diabetes mellitus
6. Neuropsychiatric disorders
7. Used bronchodilators or oral or inhaled corticosteroids in previous year

Ages: 40 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1116 (Actual)
Dates: Start 1993-09; Primary Completion 1999-05 (Actual); Study Completion 1999-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Connett, Principal Investigator — University of Minnesota

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mapp CE. Inhaled glucocorticoids in chronic obstructive pulmonary disease. N Engl J Med. 2000 Dec 28;343(26):1960-1. doi: 10.1056/NEJM200012283432609. No abstract available. PMID 11136268
- [Background] Lung Health Study Research Group; Wise R, Connett J, Weinmann G, Scanlon P, Skeans M. Effect of inhaled triamcinolone on the decline in pulmonary function in chronic obstructive pulmonary disease. N Engl J Med. 2000 Dec 28;343(26):1902-9. doi: 10.1056/NEJM200012283432601. PMID 11136260
- [Background] Simmons MS, Nides MA, Rand CS, Wise RA, Tashkin DP. Unpredictability of deception in compliance with physician-prescribed bronchodilator inhaler use in a clinical trial. Chest. 2000 Aug;118(2):290-5. doi: 10.1378/chest.118.2.290. PMID 10936115
- [Background] Tashkin DP, Murray HE, Skeans M, Murray RP. Skin manifestations of inhaled corticosteroids in COPD patients: results from Lung Health Study II. Chest. 2004 Oct;126(4):1123-33. doi: 10.1016/S0012-3692(15)31287-3. PMID 15486373
- [Background] Scanlon PD, Connett JE, Wise RA, Tashkin DP, Madhok T, Skeans M, Carpenter PC, Bailey WC, Buist AS, Eichenhorn M, Kanner RE, Weinmann G; Lung Health Study Research Group. Loss of bone density with inhaled triamcinolone in Lung Health Study II. Am J Respir Crit Care Med. 2004 Dec 15;170(12):1302-9. doi: 10.1164/rccm.200310-1349OC. Epub 2004 Sep 16. PMID 15374846
- [Background] Eichenhorn MS, Wise RA, Madhok TC, Gerald LB, Bailey WC, Tashkin DP, Scanlon PD; Lung Health Study Research Group. Lack of long-term adverse adrenal effects from inhaled triamcinolone: Lung Health Study II. Chest. 2003 Jul;124(1):57-62. doi: 10.1378/chest.124.1.57. PMID 12853502
- [Derived] Sze MA, Chen YW, Tam S, Tashkin D, Wise RA, Connett JE, Man SP, Sin DD. The relationship between Helicobacter pylori seropositivity and COPD. Thorax. 2015 Oct;70(10):923-9. doi: 10.1136/thoraxjnl-2015-207059. Epub 2015 May 29. PMID 26024688